CLINICAL TRIAL: NCT05433051
Title: A Comparison of Two Protocol for Maxillary Molar Intrusion Buccal Miniscrew and TPA Versus Vertical Holding Appliance Randomized Controlled Trial
Brief Title: A Comparison of Two Protocol for Maxillary Molar Intrusion Buccal Miniscrew and TPA Versus Vertical Holding Appliance
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mohamed Abdelrhman Shendy Abdelrhman, lecturer, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 807/220
Record Dates: First submitted 2022-06-22; First posted 2022-06-27 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Dental Intrusion; Mandibular Rotation; ANB , SNA, SNB; Openbite Teeth | Teeth and Gum | Dental
Keywords: TPA; Miniscrew; intrusion; vertical holding appliance; cephalometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Buccal miniscrews with TPA (Active Comparator): active comparator double center
  Interventions: Biological: buccal miniscrew and TPA
- vertical holding appliance (Active Comparator): active comparator double center
  Interventions: Biological: vertical holding appliance

INTERVENTIONS:
Biological: buccal miniscrew and TPA — intrusion of molars
  Arms: Buccal miniscrews with TPA
Biological: vertical holding appliance — intrusion of molars
  Arms: vertical holding appliance

SUMMARY:
this study is to compare the dental and skeletal changes caused by the intrusion of maxillary first molars buccal miniscrew and TPA versus vertical holding appliance using lateral cephalometry.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering class I or II with AOB.
* AOB ranged between 3-7 mm assessed from cephalometry.
* Patients with excess in posterior dentoalveolar height according to Burrstone .
* Patients with good oral hygiene and general health.
* Patients with no previous orthodontic treatment.
* Good quality of lateral cephalometry.

Exclusion Criteria:

* Skeletal open bite
* previous orthodontic treatment

Ages: 14 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-04-10 (Actual); Primary Completion 2024-10-10 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
amount of dental | Post-intervention at 6 months
  rate of maxillary molar intrusion by cephalometry
amount of skeletal changes | Post-intervention at 6 months
  amount of vertical overlap by cephalometry
amount of skeletal changes | Post-intervention at 6 months
  amount of mandibular rotation by cephalometry

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamed Shendy, Cairo, Nasr City, Egypt